CLINICAL TRIAL: NCT04468984
Title: Randomized, Open-Label, Phase 3 Study Evaluating Efficacy and Safety of Navitoclax in Combination With Ruxolitinib Versus Best Available Therapy in Subjects With Relapsed/Refractory Myelofibrosis (TRANSFORM-2), Incorporating Extension Arm C - Continued Access for Navitoclax to Roll Over Subjects From Studies M10-166, M16-109, M16-191, and M19-753
Brief Title: Study of Oral Navitoclax Tablet in Combination With Oral Ruxolitinib Tablet Versus Best Available Therapy to Assess Change in Spleen Volume in Adult Participants With Relapsed/Refractory Myelofibrosis
Acronym: TRANSFORM-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-178; 2023-507273-18-00 (Other: EU CT)
Expanded Access: NCT03592576 (No longer available)
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis (MF)
Keywords: ABT-263; Navitoclax; Ruxolitinib; MF; Myelofibrosis; Cancer
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms | interventions — navitoclax; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: Navitoclax + Ruxolitinib (Experimental): Participants will receive navitoclax tablets once daily and ruxolitinib tablets twice daily.
  Interventions: Drug: Navitoclax; Drug: Ruxolitinib
- Arm B: Best Available Therapy (BAT) (Active Comparator): Participants will receive one of the BAT options, per the investigator's discretion.
  Interventions: Drug: Best Available Therapy (BAT)
- Arm C: Continued Access for Navitoclax (Experimental): Participants will receive navitoclax tablets once daily.
  Interventions: Drug: Navitoclax

INTERVENTIONS:
Drug: Navitoclax — Tablet; Oral
  Arms: Arm A: Navitoclax + Ruxolitinib; Arm C: Continued Access for Navitoclax
Drug: Ruxolitinib — Tablet; Oral
  Arms: Arm A: Navitoclax + Ruxolitinib
Drug: Best Available Therapy (BAT) — Tablet/Capsule; Oral or Solution for Subcutaneous Injection
  Arms: Arm B: Best Available Therapy (BAT)

SUMMARY:
Myelofibrosis (MF) is a rare blood cancer, notable for scarring of the bone marrow (the spongy tissue inside bones) and the spleen becoming larger. The purpose of this study is to assess safety and change in spleen volume when navitoclax is given in combination with ruxolitinib, compared to best available therapy, for adult participants with MF.

Navitoclax is an investigational drug (not yet approved) being developed for the treatment of MF. Participants in this study will be randomly selected (like picking numbers out of a hat) to be in 1 of 2 treatment arms. Neither participants nor the study doctor will be able to pick which treatment arm a participants enters. In Arm A, participants will receive navitoclax in combination with ruxolitinib. In Arm B, participants will receive the best available therapy (BAT) for MF. In Arm C, participants will receive navitoclax. Adult participants with a diagnosis of MF that came back or did not get better after earlier treatment will be enrolled. Approximately 330 participants will be enrolled in approximately 322 sites across the world.

In Arm A, participants will receive navitoclax tablet by mouth once daily with by mouth ruxolitinib tablet twice daily. In Arm B, participants will receive the BAT available to the investigator. In Arm C, participants will receive navitoclax tablet by mouth once daily. Participants will receive the study drug until they experience no benefit (determined by the investigator), participants cannot tolerate the study drugs, or participants withdraw consent. The approximate treatment duration is about 3 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of treatment will be checked by medical assessments, blood and bone marrow tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must complete the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 on at least 4 out of the 7 days immediately prior to the date of randomization and must agree to collect MFSAF data daily by ePRO device during the study collection window.

  -- Has at least 2 symptoms each with an average score >= 3 or an average total score of >= 12, as measured by the MFSAF v4.0.
* Documented diagnosis of primary myelofibrosis (MF) as defined by the World Health Organization (WHO) classification, post polycythemia vera (PPV)-MF, or post essential thrombocytopenia (PET)-MF, characterized by bone marrow fibrosis grades 2 or 3.
* Classified as intermediate-2 or high-risk MF, as defined by the Dynamic International Prognostic Scoring System Plus (DIPSS+).
* Must currently be on treatment or have received prior treatment with a single Janus Kinase 2 (JAK2) inhibitor, ruxolitinib, and meet one of the following criteria (in addition to the minimum splenomegaly and symptom burden also required for eligibility):

  * Treatment with ruxolitinib for >= 24 weeks that was stopped due to lack of spleen response (refractory), or loss of spleen response or symptom control after a previous response (relapsed), or was continued despite relapsed/refractory status.
  * Treatment with ruxolitinib for < 24 weeks with documented disease progression while on therapy as defined by any of the following:

    * Appearance of new splenomegaly that is palpable to at least 5 cm below the left costal margin (LCM) in participants with no evidence of splenomegaly prior to the initiation of ruxolitinib.
    * A >= 100% increase in the palpable distance below the LCM in participants with measurable spleen distance 5 to 10 centimeters (cm) prior to the initiation of ruxolitinib.
    * A >= 50% increase in the palpable distance below the LCM in participants with measurable spleen distance > 10 cm prior to the initiation of ruxolitinib.
    * A spleen volume increase of >= 25% (as assessed by Magnetic Resonance Imaging [MRI] or Computed Tomography [CT] scan) in participants with a spleen volume assessment prior to the initiation of ruxolitinib.
  * Prior treatment with ruxolitinib of at least 10 mg twice daily (BID) for >= 28 days with intolerance defined as new RBC transfusion requirement (at least 2 units/month for 2 months) while receiving a total daily ruxolitinib dose of >= 30 mg but unable to reduce dose further due to lack of efficacy.

Note: Participant must not require a ruxolitinib dose less than 10 mg BID (20 mg daily) due to prior history of ruxolitinibrelated ≥ Grade 3 toxicity.

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Splenomegaly defined as palpable spleen measurement >= 5 cm below left costal margin or spleen volume >= 450 cm3 as assessed centrally by MRI or CT scan.
* Baseline platelet count >= 100 × 10^9/L.

Exclusion Criteria:

* Received prior treatment with a B-cell lymphoma 2 homology 3 (BH3)-mimetic compound, bromodomain and extra-terminal (BET) inhibitor, phosphoinositide 3- kinase and telomerase inhibitors (e.g., parsaclisib), prior use of > 1 JAK2 inhibitor or stem cell transplant.
* Eligible for stem cell transplantation at the time of study entry.
* Receiving medication that interferes with coagulation or platelet function within 3 days prior to the first dose of study drug or during the study treatment period except for low dose aspirin (up to 100 mg daily) and low molecular weight heparin (LMWH).
* Receiving anticancer therapy for an active malignancy or MF including chemotherapy, radiation therapy, hormonal therapy such that at least 5 half-lives of that medication is completed at least 7 days prior to the first dose of study drug or within 30 days prior to first dose of study drug, whichever is shorter, and during the study treatment period (other than any overlapping therapy as part of the selected BAT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arms A and B: Percentage of Participants who achieve Spleen Volume Reduction of at least 35% at Week 24 (SVR35W24) | At Week 24
  Reduction in spleen volume is measured by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT), per International Working Group (IWG) criteria.

SECONDARY OUTCOMES:
Arms A and B: Percentage of Participants who achieve at least 50% Reduction in Total Symptom Score (TSS) | Baseline (Week 0) Up to Week 24
  Reduction in TSS is measured by Myelofibrosis Symptom Assessment Form (MFSAF) v4.0.
Arms A and B: Percentage of Participants who achieve Spleen Volume Reduction of at least 35% at any time | Baseline (Week 0) Up to Week 97
  Reduction in spleen volume is measured by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT), per International Working Group (IWG) criteria.
Arms A and B: Percentage of Participants with Reduction in Grade of Bone Marrow Fibrosis | Baseline (Week 0) Up to Week 97
  Reduction in grade of bone marrow fibrosis from baseline as measured by the European consensus grading system will be assessed.
Arms A and B: Percentage of Participants with Anemia Response | Baseline (Week 0) Up to Week 97
  Anemia response per International Working Group (IWG) criteria will be assessed.
Arms A and B: Percentage of Participants with Overall Survival | Last Visit Up to 5 Years
  Overall survival is defined as the time from start of study to the date of death from any cause.
Arms A and B: Percentage of Participants with Leukemia-free Survival | Last Visit Up to 5 Years
  Leukemia free survival is the time from start of study to the date of development of leukemia.
Arms A and B: Percentage of Participants with Change in Fatigue | Baseline (Week 0) Up to Week 24
  Change in fatigue will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form (SF) 7a.
Arms A and B: Time to Deterioration of Physical Functioning | Baseline (Week 0) Up to Week 97
  Time to deterioration of physical functioning is measured by the physical functioning domain of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30, or death.
Arms A and B: Percentage of Participants with at Least 50% Reduction in TSS | Baseline (Week 0) Up to Week 97
  At least 50% reduction in TSS from baseline (at any time) as measured by MFSAF v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (229):
- United States (41):
  - Ironwood Cancer & Res Ctr /ID# 222162, Chandler, Arizona
  - Highlands Oncology Group, PA /ID# 221826, Springdale, Arkansas
  - City of Hope /ID# 218996, Duarte, California
  - Providence - St. Jude Medical Center /ID# 271382, Fullerton, California
  - Moores Cancer Center /ID# 271596, La Jolla, California
  - Moores Cancer Center at UC San Diego /ID# 219009, La Jolla, California
  - Long Beach Memorial Medical Ct /ID# 224542, Long Beach, California
  - Icri /Id# 221967, Whittier, California
  - St. Mary's Hospital Regional Cancer Center /ID# 224229, Grand Junction, Colorado
  - Augusta University Georgia Cancer Center /ID# 219051, Augusta, Georgia
  - Columbus Regional Research Institute /ID# 224410, Columbus, Georgia
  - University of Chicago Medical Center /ID# 271373, Chicago, Illinois
  - Northwest Oncology & Hematology - Elk Grove Village /ID# 222818, Elk Grove Village, Illinois
  - Loyola University Medical Ctr /ID# 219048, Maywood, Illinois
  - Indiana Blood & Marrow Transpl /ID# 221587, Indianapolis, Indiana
  - Tulane Medical Center - New Orleans /ID# 222940, New Orleans, Louisiana
  - Duplicate_Ochsner Clinic Foundation-New Orleans /ID# 222777, New Orleans, Louisiana
  - American Oncology Partners of Maryland /ID# 222836, Bethesda, Maryland
  - Dana-Farber Cancer Institute /ID# 218998, Boston, Massachusetts
  - University of Michigan /ID# 218463, Ann Arbor, Michigan
  - Henry Ford Hospital /ID# 221190, Detroit, Michigan
  - William Beaumont Hospital /ID# 222705, Royal Oak, Michigan
  - Saint Louis University Cancer Center /ID# 222287, St Louis, Missouri
  - Summit Medical Group-Florham Park /ID# 222620, Florham Park, New Jersey
  - Hackensack Univ Med Ctr /ID# 219047, Hackensack, New Jersey
  - The Cancer Institute at St. Francis Hospital /ID# 231782, Greenvale, New York
  - Manhattan Hematology Oncology MHO Associates /ID# 223193, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 221081, New York, New York
  - Atrium Health Wake Forest Baptist Medical Center /ID# 222899, Winston-Salem, North Carolina
  - MetroHealth Medical Center /ID# 222650, Cleveland, Ohio
  - Pennsylvania Cancer Specialists & Research Institute /ID# 271376, Gettysburg, Pennsylvania
  - Hospital of the University of Pennsylvania /ID# 219001, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center /ID# 223955, Philadelphia, Pennsylvania
  - Texas Oncology - Abilene - Antilley Road /ID# 271379, Abilene, Texas
  - Duplicate_Houston Methodist Hospital /ID# 223103, Houston, Texas
  - University of Texas Health San Antonio MD Anderson Cancer Center /ID# 233942, San Antonio, Texas
  - Utah Cancer Specialists Salt Lake Clinic /ID# 221962, Salt Lake City, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 223016, Fairfax, Virginia
  - Providence Everett /ID# 223130, Everett, Washington
  - Yakima Valley Memorial Hosp /ID# 224368, Yakima, Washington
  - HSHS St. Vincent Hospital /ID# 224468, Green Bay, Wisconsin
- Australia (5):
  - The Kinghorn Cancer Centre /ID# 221097, Darlinghurst, New South Wales
  - Border Medical Oncology Research Unit Albury Wodonga Regiona /ID# 223848, East Albury, New South Wales
  - Calvary Mater Newcastle /ID# 224324, Waratah, New South Wales
  - The Alfred Hospital /ID# 221096, Melbourne, Victoria
  - Royal Perth Hospital /ID# 221099, Perth, Western Australia
- Austria (6):
  - Universitaetsklinikum St. Poelten /ID# 221709, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 220919, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 220914, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 220915, Wels, Upper Austria
  - Medizinische Universitaet Wien /ID# 220911, Vienna, Vienna
  - Hanusch Krankenhaus /ID# 220912, Vienna
- Belgium (6):
  - ZAS Cadix /ID# 221468, Antwerp, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 224221, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Les Viviers /ID# 224827, Charleroi, Hainaut
  - UZ Gent /ID# 220841, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 228150, Sint-Niklaas, Oost-Vlaanderen
  - AZ-Delta /ID# 221469, Roeselare, West-Vlaanderen
- Bulgaria (5):
  - UMHAT Alexandrovska EAD /ID# 231652, Sofiya, Sofia
  - UMHAT Dr Georgi Stranski EAD /ID# 231650, Pleven
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 231649, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 231651, Sofia
  - UMHAT Sveta Marina /ID# 234119, Varna
- Canada (6):
  - Juravinski Cancer Centre /ID# 220887, Hamilton, Ontario
  - Ottawa Hospital Research Institute /ID# 238858, Ottawa, Ontario
  - University Health Network_Princess Margaret Cancer Centre /ID# 253942, Toronto, Ontario
  - CISSS-CA (Centre Integre de sante et de services sociaux de Chaudiere-Appalache) /ID# 222433, Lévis, Quebec
  - McGill University Health Centre - Glen Site /ID# 222614, Montreal, Quebec
  - CHUQ- Hôpital de l'Enfant-Jesus /ID# 220888, Québec, Quebec
- Croatia (5):
  - Clinical Hospital Dubrava /ID# 230801, Zagreb, City of Zagreb
  - Klinicka bolnica Merkur /ID# 230799, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 230798, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 231503, Osijek, County of Osijek-Baranja
  - Klinicki Bolnicki Centar (KBC) Split /ID# 230800, Split, Split-Dalmatia County
- Czechia (2):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 220959, Brno, Brno-mesto
  - Vseobecna fakultni nemocnice v Praze /ID# 220969, Prague
- Denmark (2):
  - Aalborg University Hospital /ID# 224391, Aalborg, North Denmark
  - Roskilde Sygehus /ID# 224456, Roskilde, Region Sjælland
- France (9):
  - Duplicate_CHU DE NICE-HOPITAL LARCHET II /ID# 256291, Nice, Alpes-Maritimes
  - CHU NIMES - Hopital Caremeau /ID# 219128, Nîmes, Gard
  - Centre Hospitalier Universitaire de Bordeaux /ID# 222696, Pessac, Gironde
  - CHU de Nantes, Hotel Dieu -HME /ID# 219127, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 222695, Pierre-Bénite, Rhone
  - Centre Hospitalier Métropole Savoie - Site Hôpital de Chambéry /ID# 223771, Chambéry, Savoie
  - Chu Angers /Id# 219129, Angers
  - Hôpital Saint-Louis /ID# 221390, Paris
  - Hopital Avicenne - APHP /ID# 221287, Bobigny, Île-de-France Region
- Germany (9):
  - Universitatsklinikum Mannheim /ID# 221529, Mannheim, Baden-Wurttemberg
  - Stauferklinikum Schwaebisch Gmuend /ID# 223948, Mutlangen, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. Heinrich und Prof. Bangerter /ID# 225025, Augsburg, Bavaria
  - Universitaetsmedizin Rostock /ID# 224157, Rostock, Mecklenburg-Vorpommern
  - Augusta-Kranken-Anstalt gGmbH, Bochum-Mitte /ID# 224695, Bochum, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH /ID# 224575, Chemnitz, Saxony
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf /ID# 221346, Dresden, Saxony
  - OncoResearch Lerchenfeld GmbH /ID# 225034, Hamburg
  - Klinikum rechts der Isar /ID# 221526, Munich
- Greece (5):
  - Olympion General Clinic /ID# 261423, Pátrai, Achaia
  - General Hospital of Athens Laiko /ID# 221175, Athens, Attica
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 221179, Athens
  - University General Hospital of Patras /ID# 221178, RION Patras Achaia
  - General Hospital of Thessaloniki George Papanikolaou /ID# 221463, Thessaloniki
- Hungary (5):
  - Fejér Vármegyei Szent György Egyetemi Oktató Kórház /ID# 220949, Székesfehérvár, Fejér
  - Debreceni Egyetem-Klinikai Kozpont /ID# 220947, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 220948, Kaposvár, Somogy County
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 220946, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Szegedi Tudományegyetem /ID# 220955, Szeged
- Israel (11):
  - Yitzhak Shamir Medical Center /ID# 222972, Ẕerifin, Central District
  - HaEmek Medical Center /ID# 220839, Afula, H_efa
  - Rambam Health Care Campus /ID# 219121, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 222973, Haifa, H_efa
  - Hadassah Medical Center-Hebrew University /ID# 219111, Jerusalem, Jerusalem
  - Hadassah Mt. Scopus /ID# 253394, Jerusalem, Jerusalem
  - Galilee Medical Center /ID# 225280, Nahariya, Northern District
  - Duplicate_Assuta Ashdod Medical Center /ID# 225281, Ashdod, Southern District
  - The Chaim Sheba Medical Center /ID# 219136, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 219135, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 219139, Petah Tikva
- Italy (15):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 221077, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Careggi /ID# 219090, Florence, Firenze
  - Duplicate_Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita /ID# 219087, Rome, Lazio
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo /ID# 225113, Monza, Monza E Brianza
  - Azienda Ospedaliera Universitaria Federico II /ID# 224673, Naples, Napoli
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 221223, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 225731, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 238438, Ancona
  - ASST Papa Giovanni XXIII /ID# 221222, Bergamo
  - AOU Policlinico G. Rodolico - San Marco /ID# 219089, Catania
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 221078, Palermo
  - Grande Ospedale Metropolitano Bianchi - Melacrino - Morelli P.O. Riuniti /ID# 221220, Reggio Calabria
  - Duplicate_University Hospital Santa Maria della Misericordia /ID# 221241, Udine
  - ASST Sette Laghi - Ospedale Di Circolo E Fondazione Macchi Varese /ID# 234183, Varese
  - Azienda ULSS 8 Berica /ID# 221079, Vicenza
- Japan (30):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 221150, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 221598, Toyoake, Aichi-ken
  - Aomori Prefectural Central Hospital /ID# 221778, Aomori, Aomori
  - Chiba University Hospital /ID# 224546, Chiba, Chiba
  - National Cancer Center Hospital East /ID# 226653, Kashiwa-shi, Chiba
  - Ehime University Hospital /ID# 221158, Toon-shi, Ehime
  - Kyushu University Hospital /ID# 221606, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 221877, Fukushima, Fukushima
  - Gifu University Hospital /ID# 224371, Gifu, Gifu
  - Sapporo Hokuyu Hospital /ID# 221149, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 221156, Kobe, Hyōgo
  - Kanazawa University Hospital /ID# 223028, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital /ID# 222044, Shiwa-gun, Iwate
  - Shonan Kamakura General Hospital /ID# 223030, Kamakura-shi, Kanagawa
  - Kumamoto Shinto General Hospital /ID# 255645, Kumamoto, Kumamoto
  - Kyoto University Hospital /ID# 223008, Kyoto, Kyoto
  - Mie University Hospital /ID# 221665, Tsu, Mie-ken
  - University of Miyazaki Hospital /ID# 221821, Miyazaki, Miyazaki
  - Niigata University Medical & Dental Hospital /ID# 223034, Niigata, Niigata
  - Kurashiki Central Hospital /ID# 221690, Kurashiki-shi, Okayama-ken
  - Kansai Medical University Hospital /ID# 257289, Hirakata-shi, Osaka
  - The University of Osaka Hospital /ID# 221159, Suita-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center /ID# 222334, Koshigaya, Saitama
  - Juntendo University Shizuoka Hospital /ID# 221780, Izunokuni-shi, Shizuoka
  - Juntendo University Hospital /ID# 221154, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 221676, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 221540, Shinjuku-ku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital /ID# 254774, Sumida-ku, Tokyo
  - University of Yamanashi Hospital /ID# 221706, Chuo-shi, Yamanashi
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo /ID# 257944, Tokyo
- Aotearoa Clinical Trials /ID# 232201, Papatoetoe, Auckland, New Zealand
- Poland (9):
  - ARS-MEDICAL Sp. z o.o. /ID# 238336, Piła, Greater Poland Voivodeship
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Medycznego im. Karola /ID# 241031, Poznan, Greater Poland Voivodeship
  - SP ZOZ Szpital Uniwersytecki w Krakowie /ID# 221160, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie /ID# 221124, Lublin, Lublin Voivodeship
  - Lux Med Onkologia - Szpital Szamocka /Id# 221265, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by Pratia /ID# 221759, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne /ID# 221298, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice /ID# 224526, Katowice
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopern /ID# 221161, Lodz, Łódź Voivodeship
- Hospital del Centro Comprensivo de Cancer de la UPR /ID# 223281, San Juan, Puerto Rico
- Russia (6):
  - Moscow State budget healthcare /ID# 221116, Moscow, Moscow
  - Clinic UZI 4D /ID# 221303, Pyatigorsk, Stavropol Kray
  - Hospital n.a. V.V. Veresaev /ID# 225221, Moscow
  - Russian Research Institute of Hematology and Transfusiology of the FMBA /ID# 221115, Saint Petersburg
  - Almazov National Medical Research Centre /ID# 221114, Saint Petersburg
  - Tula Regional Clinical Hospital /ID# 221302, Tula
- Serbia (3):
  - University Clinical Center Serbia /ID# 231058, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 231059, Belgrade, Beograd
  - University Clinical Center Vojvodina /ID# 231057, Novi Sad
- South Africa (2):
  - Duplicate_Wits Clinical Research Site /ID# 231554, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 231556, Pretoria, Gauteng
- South Korea (5):
  - Pusan National University Hospital /ID# 220980, Busan, Busan Gwang Yeogsi
  - Gachon University Gil Medical Center /ID# 220972, Incheon, Gyeonggido
  - Seoul National University Hospital /ID# 219060, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 221091, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 219061, Seoul, Seoul Teugbyeolsi
- Spain (14):
  - Complejo Hospitalario Universitario A Coruña /ID# 224617, A Coruña, A Coruna
  - Duplicate_Hospital Clínico Universitario de Santiago-CHUS /ID# 221616, Santiago de Compostela, A Coruna
  - Hospital Universitario Germans Trias i Pujol /ID# 233727, Badalona, Barcelona
  - Hospital Universitario Dr. Negrin /ID# 220923, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Central de Asturias /ID# 224815, Oviedo, Principality of Asturias
  - Hospital Parc de Salut del Mar /ID# 220922, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 240979, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 253936, Granada
  - Hospital Universitario 12 de Octubre /ID# 233726, Madrid
  - Hospital Universitario La Paz /ID# 224813, Madrid
  - Hospital Regional Universitario de Malaga /ID# 221906, Málaga
  - Hospital Universitario de Salamanca /ID# 221904, Salamanca
  - Hospital Universitario Virgen del Rocio /ID# 221932, Seville
  - Hospital Clinico Universitario de Valencia /ID# 220920, Valencia
- Skane University Hospital Lund /ID# 220834, Lund, Skåne County, Sweden
- Switzerland (2):
  - Duplicate_Universitätsspital Basel /ID# 221261, Basel, Canton of Basel-City
  - Inselspital, Universitaetsspital Bern /ID# 223439, Bern
- Taiwan (9):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 218985, Kaohsiung City, Kaohsiung
  - Chi Mei Hospital - Liouying /ID# 221144, Tainan, Tainan
  - National Taiwan University Hospital /ID# 271207, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 218980, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 271389, Kaohsiung City
  - China Medical University Hospital /ID# 218979, Taichung
  - National Cheng Kung University Hospital /ID# 271206, Tainan
  - Taipei Veterans General Hosp /ID# 221147, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 218982, Taoyuan
- Turkey (Türkiye) (7):
  - Medipol Mega Üniversite Hastanesi /ID# 271374, Tuzla, Istanbul
  - Gulhane Askeri Tip Academy /ID# 224568, Ankara
  - Hacettepe Universitesi Hastaneleri /ID# 271084, Ankara
  - Trakya University Medical Facu /ID# 224572, Edirne, Istanbul
  - Ege University Medical Faculty /ID# 224570, Izmir
  - Mersin University Medical /ID# 224571, Mersin
  - Ondokuz mayis University Facul /ID# 224567, Samsun
- Feofaniya Clinical Hospital of State Management of Affairs /ID# 271397, Kyiv, Ukraine
- United Kingdom (6):
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 221041, London, Greater London
  - United Lincolnshire Hospitals NHS Trust /ID# 224613, Lincoln, Lincolnshire
  - James Paget University Hospitals NHS Foundation Trust /ID# 221219, Great Yarmouth, Norfolk
  - University Hospitals Birmingham NHS Foundation Trust /ID# 221334, Birmingham
  - NHS Lothian /ID# 224378, Edinburgh
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 221335, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/